CLINICAL TRIAL: NCT00143000
Title: A Multicenter Study Evaluating the Efficacy and Safety of 12 Weeks Versus 24 Weeks Peginterferon Alfa-2a 40KD Combination Therapy With Ribavirin in Interferon Naïve Patients With Chronic Hepatitis C Genotype 2 or 3 Infection
Brief Title: Multicenter Study Evaluating 12 Versus 24 Weeks Therapy With Peginterferon and Ribavirin for Hepatitis C Virus (HCV) Genotype 2 or 3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NORDynamIC Study Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Swedish MPA nr. 151:2004/3458; Ethical Committee nr. Ö 763/03
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Hepatitis C Virus
Keywords: Hepatitis C Virus; Genotype 2; Genotype 3
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Peginterferon alfa-2a 40KD and Ribavirin

SUMMARY:
The primary objective of the study is to demonstrate that the efficacy of peginterferon alfa-2a 40KD combination therapy with ribavirin in interferon naïve patients with chronic hepatitis C virus infection genotype 2 or 3 given for 12 weeks is non-inferior to 24 weeks.

DETAILED DESCRIPTION:
Primary Objective of the Study: To demonstrate that the efficacy of peginterferon alfa-2a 40KD combination therapy with ribavirin in interferon naïve patients with chronic hepatitis C (CHC) virus infection genotype 2 or 3 given for 12 weeks is non-inferior to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 years of age
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Serum HCV-RNA quantifiable at >600 IU/mL by the Roche AMPLICOR HCV MONITOR® Test, v2.0.
* HCV genotype 2 or 3 infection confirmed within the past 2 years preceding the initiation of test drug dosing.
* Elevated serum ALT activity documented on at least one occasion within the past 12 months preceding the initiation of test drug dosing.
* Chronic liver disease consistent with chronic hepatitis C infection on a biopsy (obtained within the past 2 years) as judged by a local pathologist.
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Patients with cirrhosis or transition to cirrhosis must have an abdominal ultrasound, CT scan, or MRI scan without evidence of hepatocellular carcinoma and a serum AFP <100 ng/mL within 2 months of randomization
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using effective contraception during treatment and during the 6 months after treatment end

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* IFN or ribavirin therapy at any previous time
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) *6 months prior to the first dose of study drug
* Any investigational drug ≤6 weeks prior to the first dose of study drug.
* HCV genotype 1, 4, 5 or 6 infection.
* Positive test at screening for anti-HAV IgM Ab, HBsAg, anti-HBc IgM Ab, anti-HIV Ab
* Evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* History or other evidence of decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
* Serum creatinine level >2 mg/dl (>124 µmol/L) or creatinine clearance <50 ml/minute at screening
* Severe psychiatric disease, especially depression, as judged by the treating physician.
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, severe chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Thyroid dysfunction not adequately controlled (TSH and T4 levels out of normal range)
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration) or clinically relevant ophthalmological disorder due to diabetes mellitus or hypertension
* Evidence of drug abuse (including excessive alcohol consumption) in accordance with local therapeutic traditions.
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Ηemoglobin <11.3 g/dL (<7.0 mmol/L) in women or <12.9 g/dL (<8.0 mmol/L) in men at screening.
* Any patient with an increased baseline risk for anemia (e.g. thalassemia, spherocytosis, history of GI bleeding, etc) or for whom anemia would be medically problematic
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well-tolerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2004-04; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Sustained Viral Response (SVR) rate defined as percentage of patients with non-detectable HCV-RNA as measured by COBAS TaqMan 48™ (<50 IU/mL) at 24 weeks post completion of the 12 or 24 week treatment period.

SECONDARY OUTCOMES:
ALT measurements at 24 weeks post completion of the 12 or 24 week treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Norkrans, Professor, Principal Investigator — Göteborg University
Locations (1):
- Göteborg University, Gothenburg, Västra Götaland County, Sweden

REFERENCES:
- [Derived] Waldenstrom J, Hellstrand K, Westin J, Nilsson S, Christensen P, Farkkila M, Morch K, Langeland N, Norkrans G, Lagging M. Presence of interferon-lambda 4, male gender, absent/mild steatosis and low viral load augment antibody levels to hepatitis C virus. Scand J Gastroenterol. 2021 Jul;56(7):849-854. doi: 10.1080/00365521.2021.1922750. Epub 2021 Jun 2. PMID 34078234